CLINICAL TRIAL: NCT02239107
Title: N-acetyl Cysteine as an Adjuvant Therapy to Laparoscopic Ovarian Drilling in Clomiphene Citrate Resistant Polycystic Ovary Syndrome
Brief Title: N-acetyl Cysteine for Ovulation Induction in Clomiphene Citrate Resistant Polycystic Ovary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, esraa yousef badran, Esraa yousef Badran, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: n-acetyl cysteine PCOS
Record Dates: First submitted 2014-09-04; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: polycystic ovary syndrome; laparoscopic drilling; clomiphene citrate; n acetyl cysteine; insulin resistance
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-Acetyl cysteine (Experimental): Laparoscopic ovarian drilling followed by NAC 1200mg daily in two divided doses for five days starting cycle day 2 for 6 month
  Interventions: Drug: N-Acetyl cysteine; Procedure: laparoscopic ovarian drilling
- laparoscopic drilling group (Active Comparator): laparoscopic drilling only will be done
  Interventions: Procedure: laparoscopic ovarian drilling

INTERVENTIONS:
Drug: N-Acetyl cysteine
  Other Names: Acetyl cysteine; NAC
  Arms: N-Acetyl cysteine
Procedure: laparoscopic ovarian drilling

SUMMARY:
Polycystic ovary syndrome is a major endocrinological disorder affecting 5-8% of reproductive aged women. Anovulation is a major feature of the syndrome, managed primarily by clomiphene citrate. Failure to respond to clomiphene citrate is termed clomiphene resistance and second line treatment is either laparoscopic ovarian drilling or gonadotrophin ovulation induction. Although laparoscopic drilling is effective in restoring ovulation and achieving pregnancy, some women still remain anovulatory and infertile after the procedure. N-acetyl cysteine has emerged as a novel therapeutic adjuvant to laparoscopic drilling to improve ovulation and pregnancy rate.

DETAILED DESCRIPTION:
Resistance to ovulation induction therapy with clomiphene citrate (CC) is a significant problem affecting as many as 25% of patients. Laparoscopic ovarian drilling is an accepted second line treatment option, achieving ovulation in 75-90% and pregnancy in 50-69% of the CC resistant patients.

Adjuvants to laparoscopic drilling have been explored by researchers some studies have shown evidence of improved outcome with the use of N-Acetyl cystiene (NAC), a long used mucolytic drug which has been used for various other indications including detoxification and cancer chemoprotection. Several studies have addressed the possibility of using NAC as adjuvant therapy to Clomiphene citrate for induction of ovulation in resistant patients with some showing encouraging results. The use of NAC as adjuvant to laparoscopic ovarian drilling was addressed in a single pilot study showing good results with improved ovulation and pregnancy rates compared to the non users.

ELIGIBILITY:
Inclusion Criteria:

* PCOS patients according to Rotterdam criteria who failed to respond to 6 month ovulation induction therapy with clomiphene citrate,
* normal semen analysis of partner
* normal tubo-peritoneal anatomy as assessed by laparoscopy

Exclusion Criteria:

* patients who have other causes of infertility
* patients receiving gonadotrophin ovulation induction

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
ovulation rate | 6 month
  ovulation will be assessed by serial transvaginal ultrasound monitoring when feasible or day 21 serum progesterone

SECONDARY OUTCOMES:
pregnancy rate | 2 years